CLINICAL TRIAL: NCT01543516
Title: Cell Distribution in Induced Sputum in Healthy Subjects and Patients With Asthma After Different Techniques for Sputum Induction
Brief Title: Cell Distribution in Induced Sputum in Patients With Asthma
Status: Completed | Type: Observational
Sponsor: Johann Wolfgang Goethe University Hospital (Other)
Responsible Party: Principal Investigator, Dr. med. Martin Rosewich, Principal Investigator, Johann Wolfgang Goethe University Hospital
Other Study IDs: FRA-AKAS
Record Dates: First submitted 2012-02-20; First posted 2012-03-05 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Bronchial Asthma With eNO-levels Greater Than 30 ppB
Keywords: Asthma; Sputum; Blood; Inflammation; adaptive immune system; innate immune system
MeSH Terms: conditions — Asthma; Inflammation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — whole blood, serum, and sputum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with Asthma: Affected patients
  -20 Patients suffering from asthma with an eNO over 30 bbp
- Healthy Subjects: Non-affected patients
  -20 matched controls not suffering from asthma

SUMMARY:
The aim of this case-control study is the comparison of the cell distribution in induced sputum in young adults with asthma and in healthy controls.

The study consists of two visits. At both visits subjects are asked to perform a lung function test (body plethysmography) and levels of exhaled nitric oxide (eNO) are measured. At the first visit a blood sample is drawn to determine the inflammatory and allergic status of the subjects and the sputum is induced by an ultrasonic nebulizer. At the second visit another sputum sample is induced by a nozzle nebulizer. The cell distribution will be evaluated in both sputum samples.

DETAILED DESCRIPTION:
Objectives:

The aim of this study is the characterization of healthy children/ young adults and matched patients with asthma in terms of lung function, and the degree of the systemic and bronchial inflammation.

Sputum and serum samples are analyzed by quantitative real-time polymerase chain reaction (qRT-PCR) and by a cytometric bead assay (CBA). Components of the innate immune system (mannose-binding protein, TLR recognition proteins and surfactant proteins) are determined from sputum or blood respectively.

Methods and Work Programme:

This study consists of two study visits (V1 and V2)

V1 (day 0 - duration 1 hour):

* Measurement of exhaled nitric oxide (eNO)
* Lung function testing with and body plethysmography
* Blood test: blood count, CRP, RAST, serum inflammatory mediators, markers of the non-specific pulmonary defense system
* Induced sputum attained by an ultrasonic-nebulizer for inflammatory mediators and microbiological investigations

V2 (day 14-28 - duration 1 hour):

* Measurement of nitric oxide in expired air (eNO)
* Lung function testing with spirometry and body plethysmography
* Induced sputum attained by a nozzle-nebulizer for inflammatory mediators and microbiological investigations

Study population:

Children, adolescents and young people (6 - 25 years of age). Both the patients and the healthy subjects are recruited from the outpatient clinic of Pediatric Allergy and Pulmonology.

ELIGIBILITY:
Inclusion Criteria:

* informed consent
* between 6 and 25 years of age
* Known bronchial asthma/no bronchial asthma(depending on the study group)
* Ability to perform lung function tests and inhalation

Exclusion Criteria:

* < 6 and > 25 years of age
* Any acute condition with systemic or bronchial inflammation
* any chronic condition or infection (e.g. HIV, tuberculosis, malignancy)
* pregnancy
* known alcohol and/ or drug abuse
* Inability to understand the extent and scope of the study
* Participation in another study

Ages: 6 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: The study is carried out in children, adolescents, and young adults (6 to 25 years of age). Both the patients (n=20) and the healthy subjects (n=20) are recruited from the outpatient clinic of the department of Pediatric Allergy and Pulmonology, University Clinic, Goethe-University, Frankfurt/M, Germany.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2011-11; Primary Completion 2012-05 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
cell count differences in induced sputum | V1 and V2 respectively (V1 (day 0 - duration 1 hour) V2 (day 14-28 - duration 1 hour)
  Differences in neutrophils, macrophages and lymphocytes in subjects with and without asthma

SECONDARY OUTCOMES:
differences in cell count depending on the method of sputum induction | V1 and V2 respectively (V1 (day 0 - duration 1 hour) V2 (day 14-28 - duration 1 hour)
  At V1 an ultrasonic nebulizer is used for sputum induction. At V2 a breath controlled nozzle nebulizer is used for sputum induction. These different techniques might lead to different cell counts in included subjects.

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital, Goethe-University, Frankfurt am Main, Hesse, Germany

REFERENCES:
- [Derived] Koc-Gunel S, Schubert R, Zielen S, Rosewich M. Cell distribution and cytokine levels in induced sputum from healthy subjects and patients with asthma after using different nebulizer techniques. BMC Pulm Med. 2018 Jul 13;18(1):115. doi: 10.1186/s12890-018-0683-8. PMID 30005648